CLINICAL TRIAL: NCT07305051
Title: Comparison of Transhepatic and Subcostal Views for Assessing Inferior Vena Cava Diameter Variation in Cardiac Surgery Patients
Brief Title: Study Of Ultrasound Windows For Measuring Inferior Vena Cava Changes Before Cardiac Surgery
Acronym: THRIVE-CARD
Status: Not yet recruiting | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Other Study IDs: 6762
Record Dates: First submitted 2025-11-17; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-07

CONDITIONS: Perioperative Fluid Management; Hemodynamic Monitoring; Inferior Vena Cava Collapsibility Index; Cardiac Surgery Patients
Keywords: point-of-care ultrasound (POCUS); Transhepatic view; Subcostal view; Inferior vena cava (IVC); Echocardiography; Ultrasound imaging; Central venous assessment; Cardiac surgery; Fluid status assessment; Interrater reliability; Sunnybrook Health Sciences Centre; Adult patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adult Cardiac Surgery Patients: This group includes adult patients (Age ≥ 18) who are awake, spontaneously breathing, and scheduled to undergo cardiac surgery at Sunnybrook Health Sciences Centre. They must also be able to lie supine and provide informed consent.

SUMMARY:
This research study will compare two ultrasound methods for assessing the inferior vena cava (IVC), a major vein that reflects intravascular fluid status and cardiac function before and after surgery. The standard method uses a subcostal ultrasound view obtained below the breastbone, but this approach may be limited in patients with obesity, surgical dressings, or postoperative discomfort. An alternative approach, the transhepatic view, uses the liver as an acoustic window and may provide improved feasibility in these situations.

The study will evaluate whether the transhepatic view provides measurements comparable to the standard subcostal view and whether operators with different levels of ultrasound experience obtain consistent results using both methods. Adult patients who are awake and scheduled for cardiac surgery at Sunnybrook Health Sciences Centre will undergo a brief ultrasound examination before surgery. The scan takes less than 10 minutes, involves no discomfort, and does not alter clinical care. This is a minimal-risk observational study with no therapeutic interventions. Participation is voluntary, and all personal health information will remain confidential. Findings may inform future approaches to ultrasound-guided assessment and training in perioperative care.

DETAILED DESCRIPTION:
Respiratory variation in inferior vena cava (IVC) diameter is a widely accepted non-invasive marker of intravascular volume status and fluid responsiveness, particularly in spontaneously breathing patients. Among transthoracic echocardiographic windows, this variation is most commonly assessed using the subcostal (SC) view, which is considered the clinical reference standard due to its direct acoustic pathway and extensive validation in research and clinical practice. The physiologic basis for this measure is strongest in the context of spontaneous respiration, where negative intrathoracic pressure significantly influences venous return dynamics. For this reason, the study population is limited to spontaneously breathing patients to ensure physiologic consistency and interpretive validity.

The SC view, however, may be limited by factors such as body habitus, postoperative dressings, or an obstructed subxiphoid window. The transhepatic (TH) view has been proposed as a complementary or alternative approach, providing an oblique acoustic window through the liver that facilitates visualization of the IVC long axis. Several observational studies have reported strong correlation and agreement between TH and SC measurements of IVC diameter and collapsibility, including in both spontaneously breathing and mechanically ventilated patients. Despite these promising findings, prior studies have been constrained by small sample sizes, heterogeneous methodologies, and limited assessment of reproducibility-particularly across operators with different levels of ultrasound experience. These gaps underscore the need for a larger, methodologically rigorous validation study.

The primary objective of this prospective, single-center observational study is to evaluate agreement between the SC and TH views using methodological standards aligned with diagnostic accuracy frameworks such as QUADAS-2, in a larger cohort of patients scheduled for cardiac surgery. The secondary objective is to assess interrater reliability of TH and SC IVC measurements obtained by novice and expert sonographers. The results are intended to strengthen the evidence base supporting the use of the transhepatic view in perioperative care and to inform future training, competency assessment, and quality-assurance processes in point-of-care ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged eighteen years or older
* Scheduled to undergo cardiac surgery at Sunnybrook Health Sciences Centre
* Spontaneously breathing at the time of ultrasound assessment
* Able to lie supine for image acquisition
* Able to provide written informed consent

Exclusion Criteria:

* Inability to lie supine
* Known right heart failure
* Moderate to severe tricuspid regurgitation
* Portal hypertension
* End-stage renal disease
* Presence of abdominal dressings or conditions that preclude transhepatic imaging
* Poor acoustic windows that prevent adequate measurement from either the subcostal or transhepatic view, despite standard optimization techniques (positioning, breathing coaching, depth and gain adjustment, probe angulation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients scheduled to undergo elective cardiac surgery at Sunnybrook Health Sciences Centre. Eligible participants will be spontaneously breathing and able to lie supine during ultrasound assessment. The study will include male and female patients aged eighteen years or older, with no upper age limit. Exclusion criteria focus on conditions that impair accurate visualization of the inferior vena cava, including right heart failure, significant tricuspid regurgitation, portal hypertension, end-stage renal disease, obstructive dressings, or inadequate acoustic windows despite optimization maneuvers. This population reflects typical perioperative cardiac surgery patients in whom reliable non-invasive assessment of fluid status is clinically relevant.
Sampling Method: Non-Probability Sample
Enrollment: 283 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Agreement for collapsibility index (cIVC) between transhepatic and subcostal views | Preoperative period, within twenty-four to forty-eight hours before cardiac surgery.
  Outcome Metric: Intraclass correlation coefficient (ICC) for the collapsibility index (unitless).
  Rationale: To determine agreement between transhepatic and subcostal cIVC measurements.

SECONDARY OUTCOMES:
Inter-rater reliability for transhepatic collapsibility index (cIVC) | Preoperative period, during the same imaging session.
  Metric: ICC(2,1) for cIVC (unitless).
  Rationale: To assess reproducibility between novice and expert sonographers.
Agreement for IVC maximum diameter (IVCmax) | Preoperative period, during the same imaging session.
  Metrics: ICC for IVC maximum diameter (millimetres). Rationale: To determine whether transhepatic and subcostal measurements of IVC maximum diameter demonstrate sufficient agreement to support interchangeable use of the two ultrasound views for this parameter.
Bland-Altman analysis for IVC diameter ratio (IVCmax:IVCmin) | Preoperative period, during the same imaging session.
  Outcome Metric:
  Bland-Altman bias and limits of agreement for the IVC diameter ratio (unitless).
  Rationale:
  To assess systematic bias and variability in the ratio of IVC maximum to minimum diameter across the two ultrasound views, offering an additional perspective on agreement in dynamic IVC behavior.

OTHER OUTCOMES:
Agreement for IVC minimum diameter (IVCmin) | Preoperative period, during the same imaging session.
  Outcome Metric:
  Intraclass correlation coefficient (ICC) for IVC minimum diameter (millimetres).
  Rationale:
  To evaluate the agreement between transhepatic and subcostal measurements of IVC minimum diameter, which contributes to understanding the consistency of static diameter assessment across imaging windows.
Agreement for IVC diameter ratio (IVCmax:IVCmin) | Preoperative period, during the same imaging session.
  Outcome Metric:
  Intraclass correlation coefficient (ICC) for the ratio of IVC maximum to IVC minimum diameter (unitless).
  Rationale:
  To assess agreement for the proportional relationship between maximum and minimum IVC diameters, providing additional information on dynamic venous diameter behavior across ultrasound views.
Bland-Altman analysis for collapsibility index (cIVC) | Preoperative period, during the same imaging session.
  Outcome Metric:
  Bland-Altman bias and limits of agreement for the collapsibility index (unitless).
  Rationale:
  To quantify systematic bias and random variation between transhepatic and subcostal collapsibility index measurements, complementing correlation-based agreement metrics.
Bland-Altman analysis for IVC maximum diameter | Preoperative period, during the same imaging session.
  Outcome Metric:
  Bland-Altman bias and limits of agreement for IVC maximum diameter (millimeters).
  Rationale:
  To characterize systematic differences and dispersion between transhepatic and subcostal measurements of IVC maximum diameter, informing clinical interpretability of any observed discrepancies.
Bland-Altman analysis for IVC minimum diameter | Preoperative period, during the same imaging session.
  Outcome Metric:
  Bland-Altman bias and limits of agreement for IVC minimum diameter (millimeters).
  Rationale:
  To evaluate the magnitude and spread of measurement differences in IVC minimum diameter between transhepatic and subcostal views, providing a detailed assessment of potential measurement error.

CONTACTS AND LOCATIONS:
Overall Officials: Jacobo Moreno Garijo, MD, PhD, Principal Investigator — Sunnybrook Health Science Centre
Locations (1):
- Sunnybrook Health Science Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying published results (including ultrasound measurements and basic demographic variables) will be made available to qualified researchers upon reasonable request to the Principal Investigator, following publication of the primary manuscript. Data will be stored on secure institutional servers at Sunnybrook Research Institute.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: De-identified individual participant data (IPD) and supporting documents (study protocol, statistical analysis plan, and analytic code) will be made available beginning 12 months after publication of the primary manuscript. Data will remain available for a minimum of 5 years following publication, through secure institutional servers at Sunnybrook Research Institute. Access will be granted to qualified researchers upon reasonable request to the Principal Investigator, subject to a data sharing agreement that ensures privacy and appropriate use.
Access Criteria: De-identified individual participant data (IPD) and supporting documents (study protocol, statistical analysis plan, and analytic code) will be accessible to qualified researchers affiliated with academic or healthcare institutions. Requests must include a brief research proposal outlining objectives, methods, and intended use of the data. Access will be granted upon approval by the Principal Investigator and execution of a data-sharing agreement that ensures compliance with privacy, confidentiality, and ethical use standards. Approved researchers will receive access to the data through secure institutional servers at Sunnybrook Research Institute.
URL: https://sunnybrook.ca/research/

REFERENCES:
- [Background] Landis JR, Koch GG. The measurement of observer agreement for categorical data. Biometrics. 1977 Mar;33(1):159-74. PMID 843571
- [Background] Koo TK, Li MY. A Guideline of Selecting and Reporting Intraclass Correlation Coefficients for Reliability Research. J Chiropr Med. 2016 Jun;15(2):155-63. doi: 10.1016/j.jcm.2016.02.012. Epub 2016 Mar 31. PMID 27330520
- [Background] McHorney CA, Tarlov AR. Individual-patient monitoring in clinical practice: are available health status surveys adequate? Qual Life Res. 1995 Aug;4(4):293-307. doi: 10.1007/BF01593882. PMID 7550178
- [Background] Whiting PF, Rutjes AW, Westwood ME, Mallett S, Deeks JJ, Reitsma JB, Leeflang MM, Sterne JA, Bossuyt PM; QUADAS-2 Group. QUADAS-2: a revised tool for the quality assessment of diagnostic accuracy studies. Ann Intern Med. 2011 Oct 18;155(8):529-36. doi: 10.7326/0003-4819-155-8-201110180-00009. PMID 22007046
- [Background] Blehar DJ, Barton B, Gaspari RJ. Learning curves in emergency ultrasound education. Acad Emerg Med. 2015 May;22(5):574-82. doi: 10.1111/acem.12653. Epub 2015 Apr 22. PMID 25903780
- [Background] Spencer KT, Kimura BJ, Korcarz CE, Pellikka PA, Rahko PS, Siegel RJ. Focused cardiac ultrasound: recommendations from the American Society of Echocardiography. J Am Soc Echocardiogr. 2013 Jun;26(6):567-81. doi: 10.1016/j.echo.2013.04.001. No abstract available. PMID 23711341
- [Background] Sites BD, Spence BC, Gallagher JD, Wiley CW, Bertrand ML, Blike GT. Characterizing novice behavior associated with learning ultrasound-guided peripheral regional anesthesia. Reg Anesth Pain Med. 2007 Mar-Apr;32(2):107-15. doi: 10.1016/j.rapm.2006.11.006. PMID 17350520
- [Background] Croskerry P. The importance of cognitive errors in diagnosis and strategies to minimize them. Acad Med. 2003 Aug;78(8):775-80. doi: 10.1097/00001888-200308000-00003. PMID 12915363
- [Background] Sanfilippo F, La Via L, Dezio V, Santonocito C, Amelio P, Genoese G, Astuto M, Noto A. Assessment of the inferior vena cava collapsibility from subcostal and trans-hepatic imaging using both M-mode or artificial intelligence: a prospective study on healthy volunteers. Intensive Care Med Exp. 2023 Apr 3;11(1):15. doi: 10.1186/s40635-023-00505-7. PMID 37009935
- [Background] Sanfilippo F, La Via L, Dezio V, Amelio P, Genoese G, Franchi F, Messina A, Robba C, Noto A. Inferior vena cava distensibility from subcostal and trans-hepatic imaging using both M-mode or artificial intelligence: a prospective study on mechanically ventilated patients. Intensive Care Med Exp. 2023 Jul 10;11(1):40. doi: 10.1186/s40635-023-00529-z. PMID 37423948
- [Background] Hasanin A, Karam N, Mostafa M, Abdelnasser A, Hamimy W, Fouad AZ, Eladawy A, Lotfy A. THE ACCURACY OF INFERIOR VENA CAVA DISTENSIBILITY THROUGH THE TRANSHEPATIC APPROACH TO PREDICT FLUID RESPONSIVENESS IN PATIENTS WITH SEPTIC SHOCK AFTER EMERGENCY LAPAROTOMY. Shock. 2023 Oct 1;60(4):560-564. doi: 10.1097/SHK.0000000000002212. Epub 2023 Aug 23. PMID 37625114
- [Background] Bortolotti P, Colling D, Colas V, Voisin B, Dewavrin F, Poissy J, Girardie P, Kyheng M, Saulnier F, Favory R, Preau S. Respiratory changes of the inferior vena cava diameter predict fluid responsiveness in spontaneously breathing patients with cardiac arrhythmias. Ann Intensive Care. 2018 Aug 2;8(1):79. doi: 10.1186/s13613-018-0427-1. PMID 30073423
- [Background] Manzur-Sandoval D, Arteaga-Cardenas G, Gopar-Nieto R, Lazcano-Diaz E, Rojas-Velasco G. Correlation between transhepatic and subcostal inferior vena cava ultrasonographic images for evaluating fluid responsiveness after cardiac surgery. J Card Surg. 2022 Sep;37(9):2586-2591. doi: 10.1111/jocs.16696. Epub 2022 Jun 23. PMID 35735244
- [Background] Kelly N, Esteve R, Papadimos TJ, Sharpe RP, Keeney SA, DeQuevedo R, Portner M, Bahner DP, Stawicki SP. Clinician-performed ultrasound in hemodynamic and cardiac assessment: a synopsis of current indications and limitations. Eur J Trauma Emerg Surg. 2015 Oct;41(5):469-80. doi: 10.1007/s00068-014-0492-6. Epub 2015 Jan 8. PMID 26038013
- [Background] de Oliveira OH, Freitas FG, Ladeira RT, Fischer CH, Bafi AT, Azevedo LC, Machado FR. Comparison between respiratory changes in the inferior vena cava diameter and pulse pressure variation to predict fluid responsiveness in postoperative patients. J Crit Care. 2016 Aug;34:46-9. doi: 10.1016/j.jcrc.2016.03.017. Epub 2016 Mar 30. PMID 27288609
- [Background] Garijo JM, Wijeysundera DN, Munro JC, Meineri M. Correlation Between Transhepatic and Subcostal Inferior Vena Cava Views to Assess Inferior Vena Cava Variation: A Pilot Study. J Cardiothorac Vasc Anesth. 2017 Jun;31(3):973-979. doi: 10.1053/j.jvca.2017.02.003. Epub 2017 Feb 3. PMID 28366714
- [Background] Kulkarni AP, Janarthanan S, Harish MM, Suhail S, Chaudhari H, Agarwal V, Patil VP, Divatia JV. Agreement between inferior vena cava diameter measurements by subxiphoid versus transhepatic views. Indian J Crit Care Med. 2015 Dec;19(12):719-22. doi: 10.4103/0972-5229.171390. PMID 26816446
- [Background] Haroun F, Robinson M, Shayman CS, Cotton J. Subcostal versus right lateral ultrasound measurements of inferior vena cava: Measurements obtained from these two views are not equivalent in non-ICU patients. Ultrasound. 2023 Aug;31(3):196-203. doi: 10.1177/1742271X221124901. Epub 2022 Nov 16. PMID 37538967
- [Background] Ghosh S, Padhi R, Sahu S, Meher M, Jain P, Subudhi SK, Vihari J, Samal A, Sahu AK. Use of inferior vena cava guided fluid therapy in the treatment of septic shock: A randomised controlled trial. J Infect Dev Ctries. 2024 Jan 31;18(1):75-81. doi: 10.3855/jidc.18489. PMID 38377091
- [Background] Pour-Ghaz I, Manolukas T, Foray N, Raja J, Rawal A, Ibebuogu UN, Khouzam RN. Accuracy of non-invasive and minimally invasive hemodynamic monitoring: where do we stand? Ann Transl Med. 2019 Sep;7(17):421. doi: 10.21037/atm.2019.07.06. PMID 31660320
- [Background] Preau S, Bortolotti P, Colling D, Dewavrin F, Colas V, Voisin B, Onimus T, Drumez E, Durocher A, Redheuil A, Saulnier F. Diagnostic Accuracy of the Inferior Vena Cava Collapsibility to Predict Fluid Responsiveness in Spontaneously Breathing Patients With Sepsis and Acute Circulatory Failure. Crit Care Med. 2017 Mar;45(3):e290-e297. doi: 10.1097/CCM.0000000000002090. PMID 27749318
- [Background] Airapetian N, Maizel J, Alyamani O, Mahjoub Y, Lorne E, Levrard M, Ammenouche N, Seydi A, Tinturier F, Lobjoie E, Dupont H, Slama M. Does inferior vena cava respiratory variability predict fluid responsiveness in spontaneously breathing patients? Crit Care. 2015 Nov 13;19:400. doi: 10.1186/s13054-015-1100-9. PMID 26563768